CLINICAL TRIAL: NCT02068326
Title: Mentalization-Based Treatment in Groups for Adolescents With Borderline Personality Disorder (BPD) or Subthreshold BPD Versus Treatment As Usual - the M-GAB Randomized Controlled Trial
Brief Title: MBT in Groups for Adolescents With BPD or Subthreshold BPD Versus TAU - the M-GAB Randomized Controlled Trial
Acronym: M-GAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Psychiatric Research Unit, Region Zealand, Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SJ-371
Record Dates: First submitted 2014-02-19; First posted 2014-02-21 (Estimated); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Borderline Personality Disorder
Keywords: Mentalization-based Treatment; Adolescence; Borderline Personality Disorder
MeSH Terms: conditions — Borderline Personality Disorder | interventions — Mentalization-Based Therapy; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mentalization Based Treatment (Experimental): the experimental intervention is a year-long manualized program that comprises four components:
  * Five individual case-formulation sessions,
  * MBT-I, an introductory pedagogical program for patients (three weekly sessions)
  * MBT-G, MBT-program in groups (37 weekly sessions)
  * MBT-P, a psychoeducation program for the patients' parents or parents substitutes (six sessions).
  Interventions: Behavioral: Mentalization Based Treatment
- Treatment As Usual (Active Comparator): Participants randomized to the control group will receive Treatment As Usual (TAU). TAU is defined as comprising at least 12 monthly individual supportive sessions provided by non-MBT trained mental health professionals in the Department of Child and Adolescent Psychiatry in Region Zealand. Additional supportive sessions or other types of intervention may be offered to the patients according to the needs of the patients as evaluated by mental health professionals responsible for his/hers treatment. Hence, TAU may vary considerably in number and type of intervention across clinics and patients. All mental health services delivered during the treatment period to patients in the TAU group will be monitored and registered.
  Interventions: Behavioral: Treatment As Usual

INTERVENTIONS:
Behavioral: Mentalization Based Treatment
  Other Names: MBT
  Arms: Mentalization Based Treatment
Behavioral: Treatment As Usual — Treatment As Usual
  Arms: Treatment As Usual

SUMMARY:
Background: Although it is now possible to diagnose Borderline Personality Disorder (BPD) in adolescents younger than 18 years according to the Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-V), and studies indicates that BPD can be reliably diagnosed in adolescence, only a few evidence based treatment programmes for adolescent BPD exists. Mentalization-based treatment (MBT), including group psychotherapy, has repeatedly shown to be effective in treating adult BPD, but in the case of adolescents, only individual MBT have been tested and found to be effective.

Aims/hypotheses: We will test whether group based MBT (MBT-G), including an introductory programme for patients (MBT-I) and their parents (MBT-P) is more effective than Treatment As Usual (TAU) in treating adolescents with BPD or subthreshold BPD.

Methods/Design: 112 patients referred to child and adolescent psychiatric clinics in Region Zealand will be randomized to either MBT or TAU. Inclusion criteria: Meeting DSM-V BPD-criteria at the threshold (five criteria) or sub threshold level (4 criteria). Follow-up will be at three and 12 months.

Discussion: Early intervention is especially important in relation to personality psychopathology and has long-term benefits for patients, their families and society. In addition to being cost effective, using the group modality in the treatment of BPD may have several advantages. This is the first Randomized Controlled Trial (RCT) to test the effectiveness of MBT in groups for adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Meet a minimum of 4 DSM-5 BPD criteria
* Have parent's or parent substitute's commitment and ability to participate in the MBT-Parents program.
* Score 67< BPFS-C

Exclusion Criteria:

* Comorbid diagnosis of pervasive developmental disorder, learning disability (75 < IQ), anorexia, current psychosis, diagnosis of schizophrenia or schizotypal personality disorder, antisocial personality disorder as well as any other axis-I or axis-II psychopathology considered to be the primary diagnosis.
* Current psychiatric inpatient treatment
* Current (past two months) substance dependence (but not substance misuse)
* Participation in concurrent psychotherapeutic treatment outside the MBT program
* Not able to speak Danish
* Lack of informed consent

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 112 (Actual)
Dates: Start 2015-09; Primary Completion 2018-05-11 (Actual); Study Completion 2019-04-11 (Actual)

PRIMARY OUTCOMES:
The Borderline Personality Feature Scale for Children (BPFS-C) | Change from Baseline in BPFS-C at 40 weeks
The Borderline Personality Feature Scale for Children (BPFS-C) | Change from Baseline in BPFS-C at 10 weeks
The Borderline Personality Feature Scale for Children (BPFS-C) | Change from baseline at 20 weeks
The Borderline Personality Feature Scale for Children (BPFS-C) | Change from baseline at 30 weeks

SECONDARY OUTCOMES:
Becks Depression Inventory for Youth | Change from Baseline in at 10 weeks
Becks Depression Inventory for Youth | Change from Baseline in at 20 weeks
Becks Depression Inventory for Youth | Change from Baseline in at 30 weeks
Becks Depression Inventory for Youth | Change from Baseline in at 40 weeks
The Risk-Taking and Self-Harm Inventory for adolescents (RTSHIA) | Change from baseline at 40 weeks
The Risk-Taking and Self-Harm Inventory for adolescents (RTSHIA) | change from baseline at 10 weeks
The Risk-Taking and Self-Harm Inventory for adolescents (RTSHIA) | change from baseline at 20 weeks
The Risk-Taking and Self-Harm Inventory for adolescents (RTSHIA) | Chage from baseline at 30 weeks
ZAN-BPD Zanarini Rating Scale for Borderline Personality Disorder | Change from baseline at 40 weeks
The Health of the Nation Outcome Scale for Children and Adolescent (HoNOSCA) | Change from baseline at 40 weeks
The Childrens' Global Assessment Scale (CGAS) | Change from baseline at 40 weeks
The childhood behaviour checklist (CBCL, Parental outcome measure) | Change from baseline at 40 weeks
The childhood behaviour checklist (CBCL, Parental outcome measure) | Change from baseline at 10 weeks
The childhood behaviour checklist (CBCL, Parental outcome measure) | Change from baseline at 20 weeks
The childhood behaviour checklist (CBCL, Parental outcome measure) | Change from baseline at 30 weeks
The borderline personality feature scale for Children - parental version (BPFS-P) | Change from baseline at 40 weeks
The borderline personality feature scale for Children - parental version (BPFS-P) | Change from baseline at 10 weeks
The borderline personality feature scale for Children - parental version (BPFS-P) | Change from baseline at 20 weeks
The borderline personality feature scale for Children - parental version (BPFS-P) | Change from baseline at 30 weeks
Number of patients' hospital admissions and visits to the emergency room | Change from baseline at 40 weeks
The Youth Self-Report (YSR) | Change from baseline at 10 weeks
The Youth Self-Report (YSR) | Change from baseline at 20 weeks
The Youth Self-Report (YSR) | Change from baseline at 30 weeks
The Youth Self-Report (YSR) | Change from baseline at 40 weeks

OTHER OUTCOMES:
Experience of Close Relationships Inventory (ECR) | Change from baseline at 40 weeks
  Treatment related variable (mediator)
Experience of Close Relationships Inventory (ECR) | Change from baseline at 10 weeks
  Treatment related variable (mediator)
Experience of Close Relationships Inventory (ECR) | Change from baseline at 20 weeks
  Treatment related variable (mediator)
Experience of Close Relationships Inventory (ECR) | Change from baseline at 30 weeks
  Treatment related variable (mediator)
Inventory of Parent and Peer Attachment - Revised (IPPA-R) | Change from baseline at 40 weeks
  Treatment related variable (mediator)
Inventory of Parent and Peer Attachment - Revised (IPPA-R) | Change from baseline at 10 weeks
  Treatment related variable (mediator)
Inventory of Parent and Peer Attachment - Revised (IPPA-R) | Change from baseline at 20 weeks
  Treatment related variable (mediator)
Inventory of Parent and Peer Attachment - Revised (IPPA-R) | Change from baseline at 30 weeks
  Treatment related variable (mediator)
Reflective Function Questionnaire for Youth (RFQ-Y) | Change from baseline at 40 weeks
  Treatment related variable (mediator)
Reflective Function Questionnaire for Youth (RFQ-Y) | Change from baseline at 10 weeks
  Treatment related variable (mediator)
Reflective Function Questionnaire for Youth (RFQ-Y) | Change from baseline 20 weeks
  Treatment related variable (mediator)
Reflective Function Questionnaire for Youth (RFQ-Y) | Change from baseline at 30 weeks
  Treatment related variable (mediator)

CONTACTS AND LOCATIONS:
Overall Officials: Erik Simonsen, PhD, Principal Investigator — Psychiatric Research Unit, Region Zealand, Denmark
Locations (1):
- Child and Adolescent Psychiatric Department, Region Zealand, Roskilde, Region Sjælland, Denmark

REFERENCES:
- [Derived] Jorgensen MS, Storebo OJ, Bo S, Poulsen S, Gondan M, Beck E, Chanen AM, Bateman A, Pedersen J, Simonsen E. Mentalization-based treatment in groups for adolescents with Borderline Personality Disorder: 3- and 12-month follow-up of a randomized controlled trial. Eur Child Adolesc Psychiatry. 2021 May;30(5):699-710. doi: 10.1007/s00787-020-01551-2. Epub 2020 May 9. PMID 32388627
- [Derived] Storebo OJ, Stoffers-Winterling JM, Vollm BA, Kongerslev MT, Mattivi JT, Jorgensen MS, Faltinsen E, Todorovac A, Sales CP, Callesen HE, Lieb K, Simonsen E. Psychological therapies for people with borderline personality disorder. Cochrane Database Syst Rev. 2020 May 4;5(5):CD012955. doi: 10.1002/14651858.CD012955.pub2. PMID 32368793
- [Derived] Beck E, Bo S, Jorgensen MS, Gondan M, Poulsen S, Storebo OJ, Fjellerad Andersen C, Folmo E, Sharp C, Pedersen J, Simonsen E. Mentalization-based treatment in groups for adolescents with borderline personality disorder: a randomized controlled trial. J Child Psychol Psychiatry. 2020 May;61(5):594-604. doi: 10.1111/jcpp.13152. Epub 2019 Nov 8. PMID 31702058
- [Derived] Beck E, Bo S, Gondan M, Poulsen S, Pedersen L, Pedersen J, Simonsen E. Mentalization-based treatment in groups for adolescents with borderline personality disorder (BPD) or subthreshold BPD versus treatment as usual (M-GAB): study protocol for a randomized controlled trial. Trials. 2016 Jul 12;17(1):314. doi: 10.1186/s13063-016-1431-0. PMID 27405522